CLINICAL TRIAL: NCT04492124
Title: Influence of Vater's Ampulla Morphology on Biliary Cannulation Rate, Complications and Advanced Biliary Cannulation Techniques
Brief Title: Influence of Vater's Ampulla Morphology on ERCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Minho (Other)
Collaborators: Unidade Local de Saúde do Alto Minho (Other)
Responsible Party: Principal Investigator, Luis Lopes, Assistant Professor University of Minho, School of Medicine, University of Minho
Other Study IDs: 30/2020
Record Dates: First submitted 2020-07-09; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Pancreatitis
Keywords: Vater's ampulla; Major Papilla; ERCP; Biliary cannulation; Precut
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determine the influence of the papilla's morphology on the various outcomes of endoscopic retrograde cholangiopancreatography (ERCP), namely on the success of biliary cannulation, on complications, and on the need to use rescue cannulation techniques;

DETAILED DESCRIPTION:
1. Background

   ERCP is an advanced procedure which is widely used in the diagnosis and treatment of a variety of benign and malignant pancreatobiliary disorders1,2,3,4,5.

   Selective cannulation of the common bile duct (CBD) is the most important and challenging step in a biliary endoscopic retrograde cholangiopancreatography6,7. However, in the first ERCP, even in experienced hands, biliary cannulation may fail in up to 15 % - 35 % of cases when using standard methods alone8.

   Since the first description of the "Vater's papilla" by Abraham Vater in 17209, the variability in papillary morphology has been widely recognized10. The use of high quality digital images has led to a clear need and desire to create an endoscopic classification based on the papilla's morphology. During the last decade, several authors have proposed different classifications in order to predict the success of cannulation, complications and the need for more advanced cannulation techniques11,12,13,14,15. However, all the proposed classifications, with the exception of one, fail because they have not been submitted to a validation process. The only validated one is the proposed by Haraldsson13, which still has the drawback of not incorporating some of the papillary morphologies.

   Given the need, our research group created a new classification (entitled "Viana Classification") that not only incorporates more morphologies but was also validated in due course.

   Hence, the next step is to explore the potential implications of papillary morphology on the success of biliary cannulation, complications resulting from ERCP and the need to use rescue techniques (fistulotomy and double-guidewire cannulation) in the event of failure of the standard cannulation.
2. Financial resources

   All participants included in this study will perform ERCP, laboratory tests and other complementary diagnostic tests after a duly justified medical prescription (the exact same exams that the patient would do if there wasn't this study). Therefore, there are no additional costs or consumption of hospital resources.
3. Ethical considerations

   In this study, participants will be included after informed consent. Anonymity and confidentiality will be safeguarded by assigning an individual numeric code. It will also be explained the possibility of withdrawing from the study at any time, with the guarantee of the total elimination of data. All researchers involved in the study will adhere to the Rules of Ethical Conduct and Best Practices in order to comply with the precepts of the Declaration of Helsinki, the Convention on Human Rights and Biomedicine, the guidelines of the Council for International Organizations of Medical Sciences and the Guide to Good Clinical Practice.
4. Statistical analysis

   Qualitative variables will be summarized using absolute and relative frequencies, and quantitative variables will be summarized using the mean and standard deviation or the median and interquartile range, depending on their distribution profiles. The normality of the quantitative variables will be assessed using the histogram distribution.

   Relations between categorical variables will be assessed using a chi-square test and Fisher´s exact test. Differences between two or more groups of independent non-normally distributed quantitative variables will be evaluated using a Kruskal-Wallis test.

   To explain the risk of pancreatitis, a binomial logistic regression model with multiple predictors will be performed.

   The null hypothesis will be rejected when the test statistics p-values are less than <0.05. Statistical analysis, sample size calculation and graphics will be performed using Stata software (StataCorp. 2015. Stata Statistical Software: Release 14. College Station, StataCorp LP)
5. Expected results

The results from this study will contribute to a better understanding of the influence of papillary morphology on cannulation difficulty. In the event of demonstrating that some morphologies imply greater difficulty in cannulation, strategies may be created, such as the use of ab initio rescue techniques, in order to improve the results of ERCP, namely the cannulation rate.

ELIGIBILITY:
We will conduct a prospective observational study.

Inclusion Criteria:

* ERCP with indication for biliary access
* Naïve papilla

Exclusion Criteria:

* Patients unable to understand the informed consent
* Patients with surgically altered anatomy
* Patients with tumors of the papilla
* Previous sphincterotomy
* Spontaneous papillary fistula
* Papilla not visualized

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals referred for CPRE in the Digestive Endoscopy Unit of the Santa Luzia Hospital, Unidade Local de Saúde do Alto Minho, will be invited to participate in the study, in the period between June 1, 2020 to June 1, 2022.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between the morphology of the Vater's Ampulla and biliary cannulation difficulty | 1 day
  Correlation between the morphology of the Papilla de Vater, defined by the Viana classification, and the difficulty of cannulation between experts and other endoscopists (initiates and non-expert specialists)

SECONDARY OUTCOMES:
Correlation between the morphology of the Vater's Ampulla, and complications, and need/success of advanced cannulation techniques | up to 30 days
  Correlation between the morphology of the Vater's Ampulla, defined by the Viana classification, and complications, and need/success of advanced cannulation techniques (fistulotomy and double-guidewire cannulation)

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Luzia Hospital, Unidade Local de Saúde do Alto Minho, Viana do Castelo, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canena J, Liberato M, Coutinho AP, Marques I, Romao C, Veiga PM, Neves BC. Predictive value of cholangioscopy after endoscopic management of early postcholecystectomy bile duct strictures with an increasing number of plastic stents: a prospective study (with videos). Gastrointest Endosc. 2014 Feb;79(2):279-88. doi: 10.1016/j.gie.2013.07.022. Epub 2013 Sep 5. PMID 24012251
- [Background] Canena J, Coimbra J, Carvalho D, Rodrigues C, Silva M, Costa M, Horta D, Mateus Dias A, Seves I, Ramos G, Ricardo L, Coutinho AP, Romao C, Veiga PM. Endoscopic bilio-duodenal bypass: outcomes of primary and revision efficacy of combined metallic stents in malignant duodenal and biliary obstructions. Dig Dis Sci. 2014 Nov;59(11):2779-89. doi: 10.1007/s10620-014-3199-y. Epub 2014 May 13. PMID 24821464
- [Background] Canena J, Liberato M, Meireles L, Marques I, Romao C, Coutinho AP, Neves BC, Veiga PM. A non-randomized study in consecutive patients with postcholecystectomy refractory biliary leaks who were managed endoscopically with the use of multiple plastic stents or fully covered self-expandable metal stents (with videos). Gastrointest Endosc. 2015 Jul;82(1):70-8. doi: 10.1016/j.gie.2014.11.038. Epub 2015 Mar 11. PMID 25771064
- [Background] Canena J. Once upon a Time a Guideline Was Used for the Evaluation of Suspected Choledocholithiasis: A Fairy Tale or a Nightmare? GE Port J Gastroenterol. 2018 Jan;25(1):6-9. doi: 10.1159/000481688. Epub 2017 Nov 8. No abstract available. PMID 29457044
- [Background] Canena J, Lopes L, Fernandes J, Alexandrino G, Lourenco L, Libanio D, Horta D, Giestas S, Reis J. Outcomes of Single-Operator Cholangioscopy-Guided Lithotripsy in Patients with Difficult Biliary and Pancreatic Stones. GE Port J Gastroenterol. 2019 Mar;26(2):105-113. doi: 10.1159/000488508. Epub 2018 May 16. PMID 30976615
- [Background] Lopes L, Dinis-Ribeiro M, Rolanda C. Safety and efficacy of precut needle-knife fistulotomy. Scand J Gastroenterol. 2014 Jun;49(6):759-65. doi: 10.3109/00365521.2014.898085. Epub 2014 Mar 18. PMID 24641260
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Testoni PA, Testoni S, Giussani A. Difficult biliary cannulation during ERCP: how to facilitate biliary access and minimize the risk of post-ERCP pancreatitis. Dig Liver Dis. 2011 Aug;43(8):596-603. doi: 10.1016/j.dld.2011.01.019. Epub 2011 Mar 4. PMID 21377432
- [Background] Lerch MM, Domschke W. Abraham Vater of the ampulla (papilla) of Vater. Gastroenterology. 2000 Feb;118(2):379. doi: 10.1016/s0016-5085(00)70243-5. No abstract available. PMID 10691372
- [Background] Vater A. Dissertatio anatomica quo novum bilis dicetilicum circa orifucum ductus choledochi ut et valvulosam colli vesicæ felleæ constructionem ad disceptandum proponit. Wittenberg 1720
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N. Effect of precut sphincterotomy on biliary cannulation based on the characteristics of the major duodenal papilla. Clin Gastroenterol Hepatol. 2007 Sep;5(9):1113-8. doi: 10.1016/j.cgh.2007.05.014. Epub 2007 Aug 6. PMID 17689295
- [Background] Lee TH, Bang BW, Park SH, Jeong S, Lee DH, Kim SJ. Precut fistulotomy for difficult biliary cannulation: is it a risky preference in relation to the experience of an endoscopist? Dig Dis Sci. 2011 Jun;56(6):1896-903. doi: 10.1007/s10620-010-1483-z. Epub 2010 Nov 17. PMID 21082346
- [Background] Haraldsson E, Lundell L, Swahn F, Enochsson L, Lohr JM, Arnelo U; Scandinavian Association for Digestive Endoscopy (SADE) Study Group of Endoscopic Retrograde Cholangio-Pancreaticography. Endoscopic classification of the papilla of Vater. Results of an inter- and intraobserver agreement study. United European Gastroenterol J. 2017 Jun;5(4):504-510. doi: 10.1177/2050640616674837. Epub 2016 Oct 17. PMID 28588881
- [Background] Haraldsson E, Kylanpaa L, Gronroos J, Saarela A, Toth E, Qvigstad G, Hult M, Lindstrom O, Laine S, Karjula H, Hauge T, Sadik R, Arnelo U. Macroscopic appearance of the major duodenal papilla influences bile duct cannulation: a prospective multicenter study by the Scandinavian Association for Digestive Endoscopy Study Group for ERCP. Gastrointest Endosc. 2019 Dec;90(6):957-963. doi: 10.1016/j.gie.2019.07.014. Epub 2019 Jul 18. PMID 31326385
- [Background] Watanabe M, Okuwaki K, Kida M, Imaizumi H, Yamauchi H, Kaneko T, Iwai T, Hasegawa R, Miyata E, Masutani H, Tadehara M, Adachi K, Koizumi W. Transpapillary Biliary Cannulation is Difficult in Cases with Large Oral Protrusion of the Duodenal Papilla. Dig Dis Sci. 2019 Aug;64(8):2291-2299. doi: 10.1007/s10620-019-05510-z. Epub 2019 Feb 12. PMID 30746630